CLINICAL TRIAL: NCT03929406
Title: Stimulation cérébrale Profonde et Empreinte Tissulaire : Une Nouvelle stratégie Pour la Recherche Biologique in Vivo Dans la Maladie de Parkinson, Les TOC, la Dystonie, le Tremblement Essentiel et le Syndrome Gilles de la Tourette.
Brief Title: Brain Tissue Imprint
Acronym: BTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A03001-54
Record Dates: First submitted 2019-04-09; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-03

CONDITIONS: Parkinson Disease; Neurologic Disorder
Keywords: Deep Brain Stimulation; Tissue harvesting; Molecular analysis - Proteomics
MeSH Terms: conditions — Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Tissue Imprint (Experimental): Evaluation and validation of the samples collected during the brain tissue imprint procedure using a CE marked Medical Device in patients presenting one of the following five disorders: Parkinson's disease (PD), essential tremor (ET), dystonia (DYS), Obsessive compulsive disorder (OCD) and Tourette Syndrome (TS).
  Interventions: Device: Brain Tissue Imprint

INTERVENTIONS:
Device: Brain Tissue Imprint — Brain Tissue Imprint procedure (BTI) is performed during DBS surgery. Before the implantation of the electrode, the surgeon uses a dilator. It is a rigid stylet with a blunt end, intended to prepare the way for the final electrode. This dilator is lowered gently through the cerebral parenchyma up to the target then removed to be replaced by the electrode.
  In our BTI study, the standard dilator used in DBS surgery will be replaced by a CE marked Medical Device. This brain imprint kit will be used for each hemisphere. The procedure is the following:
  * The guide tube with the first stylet is set up to the target
  * Withdrawal of the first stylet and insertion of the second stylet for one minute to have a spontaneous and adequate tissue adhesion
  * Withdrawal of the guide tube containing the stylet. This last step will prevent contamination of the harvested material on the stylet during the removal.

SUMMARY:
This exploratory study aims to validate the collection and analysis of brain tissue imprints during the DBS by using a CE marked Medical Device in patients presenting one of the following five disorders: Parkinson's disease (PD), essential tremor (ET), dystonia (DYS), Obsessive compulsive disorder (OCD) and Tourette Syndrome (TS).

The Brain Tissue Imprint project is focused on the DBS surgical procedure, which constitutes an appropriate method to collect brain tissue imprints by taking advantage of the direct and transitory contact at the extremity of the dilator with adjacent brain tissue. Indeed, during this step, micro-fragments of brain material spontaneously adhere to the dilator tip. It is this imprinting process that allows to collect what is defined as "brain tissue imprints. This approach is part of the standard surgical procedure of the SCP without major change or complications.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) has become the standard functional neurosurgery treatment for drug resistant Parkinson's disease (PD) patients. It has also demonstrated its efficacy to treat various movement disorders as well as neurological and psychiatric disorders. The subthalamic nucleus (STN), the globus pallidus internal (GPi) or the ventral intermediate nucleus of the thalamus (VIM) are the major targets of DBS.

Access to pathological brain tissue in living PD patients or other neurological diseases is a key issue for the discovery of new therapeutic targets and the development of potential curative therapies. In this context, DBS offers a unique access to the pathological brain. In the standard surgical procedure, to prepare the way for the final electrode, the surgeon uses a dilator that is lowered gently through the cerebral parenchyma up to the target. It has been shown that during this step, brain tissue fragments adhere to the extremity of the dilator. However, the major drawback of the standard dilator lies in the fact that its end is in contact with several brain regions before reaching the targeted nucleus. Therefore, it is difficult to guarantee the origin of the collected tissue micro-fragments. In order to optimize the specificity of the harvested imprints, the investgator will use a dedicated CE marked medical device that consists of a guide tube and a stylet instead of the dilator used in DBS surgical procedure. The objective of this study is to validate brain tissue imprints collection in PD, ET, DYS, OCD and TS.

The BTI will be specifically collected from the targeted implantation site corresponding to the STN, the GPi and the VIM. Moreover, the tip of the electrode (and therefore the BTI) often reaches the substantia negra pars compacta (SNpc) because of its proximity with the STN. The ability to perform BTI in the SNpc is of highly interest since it is the structure containing the neurons that degenerate gradually and massively throughout the pathological process of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients for deep brain stimulation surgery
* Patients affiliated to social security or benefiting of a similar insurance scheme
* Patients having signed a consent to participate to the study

Exclusion Criteria:

* Patient not eligible for deep brain stimulation surgery
* Pregnant women or nursing mothers
* Persons deprived of liberty by judicial or administrative decision
* Persons unable to express their consent or legally protected
* Persons in period of disqualification for another interventional research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Validation of the collection of brain tissue fragments on the BTI device during the DBS surgical procedure | The evaluation of the collection of brain tissue fragments will be performed in the surgery room when the BTI device is removed from the patient and inserted in the collection tube
  Visual assessment of the presence or the absence of a tissue micro-fragment. The presence or absence of blood contamination will also be notified

CONTACTS AND LOCATIONS:
Overall Officials: Stéphan Chabardès, Pr, Principal Investigator — Grenoble Hospital - Service de Neurochirurgie, CHUGA
Locations (1):
- Grenoble Hospital - CHUGA, Grenoble, Isere, France

REFERENCES:
- [Background] Benabid AL, Pollak P, Louveau A, Henry S, de Rougemont J. Combined (thalamotomy and stimulation) stereotactic surgery of the VIM thalamic nucleus for bilateral Parkinson disease. Appl Neurophysiol. 1987;50(1-6):344-6. doi: 10.1159/000100803. PMID 3329873
- [Background] Perlmutter JS, Mink JW. Deep brain stimulation. Annu Rev Neurosci. 2006;29:229-57. doi: 10.1146/annurev.neuro.29.051605.112824. PMID 16776585
- [Background] Holtzheimer PE, Mayberg HS. Deep brain stimulation for psychiatric disorders. Annu Rev Neurosci. 2011;34:289-307. doi: 10.1146/annurev-neuro-061010-113638. PMID 21692660
- [Background] Hariz M, Blomstedt P, Zrinzo L. Future of brain stimulation: new targets, new indications, new technology. Mov Disord. 2013 Nov;28(13):1784-92. doi: 10.1002/mds.25665. Epub 2013 Oct 7. PMID 24123327
- [Background] Fontaine D, Lanteri-Minet M, Ouchchane L, Lazorthes Y, Mertens P, Blond S, Geraud G, Fabre N, Navez M, Lucas C, Dubois F, Sol JC, Paquis P, Lemaire JJ. Anatomical location of effective deep brain stimulation electrodes in chronic cluster headache. Brain. 2010 Apr;133(Pt 4):1214-23. doi: 10.1093/brain/awq041. Epub 2010 Mar 17. PMID 20237130
- [Background] Laxton AW, Tang-Wai DF, McAndrews MP, Zumsteg D, Wennberg R, Keren R, Wherrett J, Naglie G, Hamani C, Smith GS, Lozano AM. A phase I trial of deep brain stimulation of memory circuits in Alzheimer's disease. Ann Neurol. 2010 Oct;68(4):521-34. doi: 10.1002/ana.22089. PMID 20687206
- [Background] Boex C, Seeck M, Vulliemoz S, Rossetti AO, Staedler C, Spinelli L, Pegna AJ, Pralong E, Villemure JG, Foletti G, Pollo C. Chronic deep brain stimulation in mesial temporal lobe epilepsy. Seizure. 2011 Jul;20(6):485-90. doi: 10.1016/j.seizure.2011.03.001. Epub 2011 Apr 12. PMID 21489828
- [Background] Lozano AM, Giacobbe P, Hamani C, Rizvi SJ, Kennedy SH, Kolivakis TT, Debonnel G, Sadikot AF, Lam RW, Howard AK, Ilcewicz-Klimek M, Honey CR, Mayberg HS. A multicenter pilot study of subcallosal cingulate area deep brain stimulation for treatment-resistant depression. J Neurosurg. 2012 Feb;116(2):315-22. doi: 10.3171/2011.10.JNS102122. Epub 2011 Nov 18. PMID 22098195
- [Background] Torres N, Chabardes S, Piallat B, Devergnas A, Benabid AL. Body fat and body weight reduction following hypothalamic deep brain stimulation in monkeys: an intraventricular approach. Int J Obes (Lond). 2012 Dec;36(12):1537-44. doi: 10.1038/ijo.2011.271. Epub 2012 Feb 21. PMID 22349575
- [Background] Luigjes J, van den Brink W, Feenstra M, van den Munckhof P, Schuurman PR, Schippers R, Mazaheri A, De Vries TJ, Denys D. Deep brain stimulation in addiction: a review of potential brain targets. Mol Psychiatry. 2012 Jun;17(6):572-83. doi: 10.1038/mp.2011.114. Epub 2011 Sep 20. PMID 21931318
- [Background] Benabid AL, Chabardes S, Mitrofanis J, Pollak P. Deep brain stimulation of the subthalamic nucleus for the treatment of Parkinson's disease. Lancet Neurol. 2009 Jan;8(1):67-81. doi: 10.1016/S1474-4422(08)70291-6. PMID 19081516
- [Background] Zaccaria A, Bouamrani A, Chabardes S, El Atifi M, Seigneuret E, Lobrinus JA, Dubois-Dauphin M, Berger F, Burkhard PR. Deep brain stimulation-associated brain tissue imprints: a new in vivo approach to biological research in human Parkinson's disease. Mol Neurodegener. 2016 Jan 28;11:12. doi: 10.1186/s13024-016-0077-4. PMID 26822202
- [Background] Crecelius A, Gotz A, Arzberger T, Frohlich T, Arnold GJ, Ferrer I, Kretzschmar HA. Assessing quantitative post-mortem changes in the gray matter of the human frontal cortex proteome by 2-D DIGE. Proteomics. 2008 Mar;8(6):1276-91. doi: 10.1002/pmic.200700728. PMID 18283663
- [Background] Mexal S, Berger R, Adams CE, Ross RG, Freedman R, Leonard S. Brain pH has a significant impact on human postmortem hippocampal gene expression profiles. Brain Res. 2006 Aug 23;1106(1):1-11. doi: 10.1016/j.brainres.2006.05.043. Epub 2006 Jul 14. PMID 16843448
- [Background] Chariot P, Witt K, Pautot V, Porcher R, Thomas G, Zafrani ES, Lemaire F. Declining autopsy rate in a French hospital: physician's attitudes to the autopsy and use of autopsy material in research publications. Arch Pathol Lab Med. 2000 May;124(5):739-45. doi: 10.5858/2000-124-0739-DARIAF. PMID 10782159